CLINICAL TRIAL: NCT02320942
Title: Implementation of a Physician-prescribed Exercise Program as Standard of Care in Allogeneic Stem Cell Transplant Patients in British Columbia: a Pilot Study.
Brief Title: Exercise Post Bone Marrow Transplant
Acronym: ExP-BMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H14-01679
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Leukemia
Keywords: Bone Marrow Transplantation; Exercise; Rehabilitation; Cancer
MeSH Terms: conditions — Leukemia; Motor Activity; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise Intervention (Experimental): At discharge from the inpatient unit, participants will receive a practical introduction by an exercise specialist and enrolled in the 12-week exercise intervention
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Exercise Intervention — The semi-supervised intervention is a progressive program with a goal of three aerobic and two resistance exercise sessions per week. Aerobic exercise will consist of 20-40 minutes of bicycling using a stationary bike located on CP6 (supervised or un-supervised) or brisk walking at home. Resistance exercise will include exercise for the upper and lower extremities with stretch bands. Patients will complete at least one supervised aerobic and resistance session per week with the exercise trainer and complete a daily log of their exercise, including adherence, adverse events and symptoms.

SUMMARY:
This study is a preliminary study to assess whether it is possible to introduce an exercise program for BMT patients after discharge from hospital. The exercise program will include 3 endurance (stationary bike, walking) and 2 resistance (weights, stretch bands) training sessions/week, until 100 days after BMT. Our second plan is to test changes in QoL, aerobic fitness, muscle strength, total body fat and mineral composition, and blood immune markers with exercise in the 100 days after BMT. The investigators anticipate this study will improve the QoL, mobility, and strength of patients after BMT, therefore allowing a faster and healthier recovery.

DETAILED DESCRIPTION:
PURPOSE: Our long-term goal is to conduct a randomized clinical trial to investigate whether a physician-prescribed supervised exercise intervention in allogeneic stem cell transplant (alloHSCT) patients within the Leukemia/Bone Marrow Transplant (LBMT) Program of BC results in improved QoL compared to no intervention. This current study is a pilot study with the primary aim of determining the feasibility, including recruitment, retention, and adherence, of delivering such an intervention as standard of care.

HYPOTHESES:

1. The physician-prescribed exercise intervention will be feasible in terms of recruitment (goal of 20 patients recruited over study period), retention (≥70%), and adherence (≥70%) of participants.
2. The intervention will be safe and highly acceptable to participants.

JUSTIFICATION: Allogeneic hematopoeitic stem cell transplantation (alloHSCT) is used to treat malignant and non-malignant hematopoeitic diseases including leukemia, lymphoma, and bone marrow failure syndromes. Recent advances in alloHSCT have led to improved relapse-free and overall survival (OS); however alloHSCT remains associated with significant morbidity including chronic graft-versus-host disease (GVHD), infectious and immune complications, reduced physical performance and functioning due to deconditioning, sarcopenia, and bone loss, and particularly high levels of fatigue and psycho-social stress, all of which negatively impact patients' quality of life (QoL). There is an accumulating body of evidence emphasizing that physical activity (PA) may be one modifiable lifestyle factor that has the potential to positively influence QoL, physical functioning and other health-related outcomes in HSCT survivors. Currently alloHSCT patients in Canada, including in BC, have little access to exercise programs that address the unique barriers within this population, particularly during the early post-transplant period where the need is greatest. These include concerns about using a public gym due to an immunocompromised state, supervision by trained professionals, and ability to exercise with low blood counts and other post-transplant complications.

OBJECTIVES:

1. To determine the feasibility (recruitment, retention, and adherence) of delivering a physician-prescribed supervised exercise intervention in alloHSCT recipients as standard of care.
2. To assess changes in health-related quality of life (HRQoL), fatigue, physical functioning, body composition, biomarkers of immune reconstitution, and therapy-related toxicity with the institution of a physician-prescribed supervised exercise intervention in alloHSCT recipients.

RESEARCH METHOD:

Study Design and Population: This study is a prospective pre-post test single-arm pilot study to assess the feasibility of the intervention. Eligible participants are adults ≥ 18 years of age undergoing alloHSCT for any indication through the LBMT Program of BC at VGH. Participants must be able to fill out questionnaires in English. Participants will be excluded if they have contraindications to entrance into an exercise program (i.e., musculoskeletal issue or not cleared for exercise by the attending physician). Eligible participants will be identified by their transplant physicians and informed consent will be obtained by the research team.

Intervention: At discharge from the inpatient unit, participants will receive a practical introduction by an exercise specialist and enrolled in the 12-week exercise intervention. The semi-supervised intervention is a progressive program with a goal of three aerobic and two resistance exercise sessions per week. Aerobic exercise will consist of 20-40 minutes of bicycling using a stationary bike located on CP6 (supervised or un-supervised) or brisk walking at home. Resistance exercise will include exercise for the upper and lower extremities with stretch bands (8-20 repetitions, 2 or 3 sets). Patients will complete at least one supervised aerobic and resistance session per week with the exercise trainer and complete a daily log of their exercise, including adherence, adverse events and symptoms. At the weekly supervised session, the exercise specialist will review adherence to the intervention and provide support for questions and overcoming identified barriers to adherence. Contraindications for starting a training session will include active infection (temperature > 38oC), severe pain, nausea and dizziness, platelet counts < 20 000/uL and Hb < 80 g/L. Exercise sessions will be stopped if pain, dizziness, or other contraindications occur. These contraindications are in keeping with previous studies of exercise in this population that have been deemed safe.

Data Collection and Endpoints: Follow-up assessments will occur at baseline (pre-BMT visit), on discharge from the inpatient ward (within the first week of attending CP6), day 60, and day 100 post-BMT (approximately 12-weeks).

Baseline demographics: Demographic data will be collected by patient interviews at baseline, including age, other health conditions and physical activity levels prior to HSCT. Medical and transplantation variables will be obtained from patients' medical records.

HRQoL: Patients QoL will be assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30), which evaluates different factors of HRQoL in 5 functional and 9 symptom subscales/items, as well as a global score of HRQoL. This tool has been used extensively in the HSCT population, including in 6 of the 7 trials identified in our systematic review and meta-analysis of exercise effects on HRQoL in HSCT patients.

Functional assessment: PFTs will be done at baseline and day 100 as is already standard of care. Aerobic fitness will be assessed using the 6 minute walk test (6MWT) protocol by the American Thoracic Society. This test has been used extensively in clinical exercise trials to estimate aerobic capacity and has been tested in the HSCT population. Muscle strength will be evaluated by the 30-second chair stand (lower extremity), which is a component of the Senior's Fitness test, and grip strength (upper extremity). Mobility will be measured by the time-up-and go test. This testing will be completed on CP6 by the exercise specialist.

Body Composition Analysis: Standing height, body weight, and waist and hip circumferences will be measured. Baseline bone mineral density testing (BMD), 1,25-OH vitamin D and calcium levels, and dual-energy X-ray absorptiometry (DXA) scan are performed by Dr. Kendler, pre-transplant and at day +100 as standard of care. The DXA scan is a well validated tool which accurately and precisely measures lean, fat, and mineral composition and has a number of strengths compared to other modalities of body composition measurement.

Immune function: Markers of immune function including total white blood cell count, lymphocyte count, CD4+ and CD8+ subsets of T-lymphocytes, and T-regulatory cells will be tested pre-BMT and at Day 100. These markers have been previously evaluated in studies of exercise interventions in HSCT patients with inconsistent results.

STATISTICAL ANALYSIS

Primary Aim (Objective 1): For the larger RCT, sample size is based on an expected mean change in global HRQoL in the intervention group of 5 points and standard deviations from the literature based on prior studies using the EORTC-QLQ-C30 questionnaire. We would be able to reject the null hypothesis that the mean change in global HRQoL between the intervention and control groups are equal with a power of 80% if we enroll 41 patients in each group. The Type I error probability associated with this test of this null hypothesis is 0.05 and is two-sided. To account for a maximum 30% dropout rate (based on an expected 20% transplant-related mortality and 10% dropout rate), we plan to enroll 120 patients (60 in each group) in the larger RCT. This may be modified based on the results of the current study. Specific feasibility objectives of this study are:

1. To determine study recruitment rates: The study will be considered feasible if we recruit 20 participants. Over the last 5 years, the average number of alloHSCTs performed at VGH through the LBMT Program of BC was 90 per year, which averages to approximately 30 transplants per 4-month period. Based on a preparatory period of 2 months, recruitment over a 4-month period, the requirement for 100 days (3-4 months) follow-up from the last patient enrolled, and time for analyses (see Project Timeline), 20 patients is a reasonable recruitment target for this pilot study. This translates into 20 patients per 4-month period, which would mean a minimum of 2 years to recruit 120 patients for the larger trial. Recruitment rate will be assessed at an interim mark of 2 months. If below anticipated, we will review with our team the barriers to recruitment and modify recruiting strategy.
2. To determine study retention rates: This study will be considered feasible if ≥ 70% of the sample complete the day 100 assessment. Prior studies have demonstrated that 72%38 and 77%40 of patients complete the final assessment, forming the basis of our estimate.
3. To determine adherence of the exercise intervention: The intervention will be considered feasible if participants complete ≥ 70% of the prescribed number of exercise sessions at the end of the follow-up. Prior data indicate that adherence to PA interventions in alloHSCT patients is 85%, ranging from 68% to 90%.24 We have reduced to 70% due to the medical acuity of the participants and possible competing time demands of active medical treatments.
4. Recruitment and retention will be summarized using a CONSORT flow diagram (http://www.consort-statement.org/). Analysis of the feasibility objectives will be descriptive or based on estimates with 95% confidence intervals.

Secondary Aim (Objective 2): Descriptive statistics will be reported as means and standard deviations for continuous variables and number (%) for categorical variables. Changes in outcome variables from baseline to day 100 will be analyzed using a paired-samples t test (continuous data), Wilcoxon signed ranks test (ordinal data), or McNemar's test (categorical data). For variables also assessed at discharge and day 60, a repeated measures analysis of variance will be used. Subgroup analyses will be conducted for patients based on intensity of conditioning regimen (myeloablative versus reduced-intensity) and based on whether or not patients receive glucocorticoid therapy. Statistical analysis will be performed using STATA version 12.1 (College Station, TX) and a type I error rate of 0.05 will be assumed for all statistical tests. The Bonferroni method will be used to adjust the level of significance for multiple testing of secondary outcomes so the overall level is alpha=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Undergoing alloHSCT for any indication through the LBMT Program of BC at VGH
* Good comprehension of English (must be able to fill out questionnaires in English)

Exclusion Criteria:

* Contraindications to entrance into an exercise program (i.e., known cardiovascular disease, musculoskeletal issue or not cleared for exercise by the attending physician)
* Mobility impairment requiring use of mobility aids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | Approximately 12-weeks
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30).

SECONDARY OUTCOMES:
Baseline Demographics | Baseline: pre-BMT visit.
  Demographic data will be collected by patient interviews at baseline, including age, other health conditions and physical activity levels prior to HSCT. Medical and transplantation variables will be obtained from patients' medical records.
Aerobic Fitness | Approximately 12-weeks
  Aerobic fitness will be assessed using the 6 minute walk test (6MWT) protocol by the American Thoracic Society. This test has been used extensively in clinical exercise trials to estimate aerobic capacity and has been tested in the HSCT population.
Muscle Strength | Approximately 12-weeks
  Muscle strength will be evaluated by the 30-second chair stand (lower extremity), which is a component of the Senior's Fitness test, and grip strength (upper extremity). Mobility will be measured by the time-up-and go test.
Body Composition | Approximately 12-weeks
  Standing height, body weight, and waist and hip circumferences will be measured. Baseline bone mineral density testing (BMD), 1,25-OH vitamin D and calcium levels, and dual-energy X-ray absorptiometry (DXA) scan are performed by Dr. Kendler, pre-transplant and at day +100 as standard of care. The DXA scan is a well validated tool which accurately and precisely measures lean, fat, and mineral composition and has a number of strengths compared to other modalities of body composition measurement.
Immune Function | Approximately 12-weeks
  Markers of immune function including total white blood cell count, lymphocyte count, CD4+ and CD8+ subsets of T-lymphocytes, and T-regulatory cells will be tested pre-BMT and at Day 100. These markers have been previously evaluated in studies of exercise interventions in HSCT patients with inconsistent results.

CONTACTS AND LOCATIONS:
Overall Officials: Raewyn Broady, MBChB, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- Vancouver General Hospital - Krall Centre Centennial Pavilion 6, Vancouver, British Columbia, Canada